CLINICAL TRIAL: NCT05989100
Title: Effects of Taste Stimulation on Swallowing Function of Patient With Post-stroke Dysphagia and Its Mechanism
Brief Title: Taste Stimulation for Post-stroke Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KYLL-202307-024
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Dysphagia
Keywords: taste stimulation; sour stimulaiton; thermal stimulation; functional near-inrared spectroscopy
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Favourate taste stimulation group, sour stimulation group and thermal stimulation group.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Favourate taste stimulation (Experimental): The swab will be immersed in sugar, salt, citric acid, or paprika mixed with water, and be placed in -18℃ refrigerator. Select the swabs of the participant favourate taste to brush oral cavity and tounge. The stimulation will last two to three minutes one time, and twice for a rehabilitation session, once per day and six days every week, three weeks totally. Swallowing rehabilitation also include standard training that carried out in the department.
  Interventions: Behavioral: Favourate taste stimulation
- Sour stimulation (Active Comparator): Using sour swab to brush oral cavity and tounge of the participant. The treatment duration and other training method is as same as mentioned above.
  Interventions: Behavioral: Sour taste stimulation
- Thermal stimulation (Placebo Comparator): Only ice-water swab to brush oral cavity and tounge. The treatment duration and other training method is as same as mentioned above.
  Interventions: Behavioral: Thermal stimulation group

INTERVENTIONS:
Behavioral: Favourate taste stimulation — The taste stimulaiton for swallowing is completed with long swab. Taste solution will be prepared with sugar, salt, citric acid, or paprika mixed with water. And the swab will be immersed in the solution and freezed in -18℃ circumstances. Bilateral buccal mucosa，palate and tounge will be brushed. Four swabs will be used in a training session.
  Arms: Favourate taste stimulation
Behavioral: Sour taste stimulation — Using sour swab to brush oral cavity and tounge.
  Arms: Sour stimulation
Behavioral: Thermal stimulation group — Only ice-water swab to brush oral cavity and tounge.
  Arms: Thermal stimulation

SUMMARY:
The goal of this clinical study is to compare the effect of favourate taste stimulation of oral cavity and tounge, with sour and traditional single thermal stimulation in post-stroke patients with dysphagia. The main questions it aims to answer are:

1. Whether favourate taste stimulation of oral and tounge is better than traditional thermal stimulation in improving swallowing function of patients with dysphagia.
2. It has been reported that taste of sour stimulation can increase the frequency of swallowing. In this study, we want to know which is better for improving swallowing function between favourate taste stimulation and sour taste stimulation.
3. Functional near-infrared spectroscopy (fNIRS) will be applied in this study to understand the neural mechanism of taste stimulation in improving swallowing function.

Participants screened as post-stroke dysphagia will accept swallowing evaluation and fNIRS test before and after treatment. The treatment include taste stimulation and traditional swallowing training.

Researchers will compare favourate taste stimulation with sour-taste stimulation and single thermal stimulation to see if the swallowing function improved faster and better in favourate taste stimulation group.

DETAILED DESCRIPTION:
Taste perception can help to initiate swallow. Different taste has different impact on swallowing function. Patients with post-stroke dysphagia always have taste impairment and initiation delay of swallowing. In this study, patients with dysphagia after stroke will be recruited and treated with favourate taste stimulation or sour taste stimulation or non-taste stimulation for 2 weeks. Traditional swallowing rehabilitation will be applied base on the status of patients. Before and after the treatment, participants completed swallowing assessment, including quantitative measurement of hyoid displacement, functional oral intake scale (FOIS), dysphagia severity rating scale (DSRS), and standardized swallowing assessment (SSA). In order to understand the effect of taste stimulation on brain network, fNIRS will be conducted.The participants have to conduct these examination three to four weeks after the treatment to undertand the long-time effect of taste stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as first-ever stroke and diagnosed as dysphagia with modified water swallowing test, duration of dysphagia was more than one month;
2. can complete all the test with MMSE >15;
3. agree to participate the experiment, and sign the written informed consent.

Exclusion Criteria:

1. have other diseases that could induce dysphagia, such as cranial and neck tumor, history of radiotherapy or chemotherapy, tongue muscle atrophy, myasthenia gravis, parotid tumor and multiple sclerosis, etc;
2. lose of taste perception;
3. combined with other major disease that can not tolerate the examination and swallowing training;
4. surgery of cranial allogeneic plasticity, scalp ulcer or damage that thought as contraindications of fNIRS.
5. with other neurological conditions (eg, Parkinson's disease, dementia).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Hyoid displacement | Befor and after the three-week treatment, and 3 weeks after the treatment.
  The probe of ultrosound will be placed in the middle of the neck, paralled to the sagittal line. Record the video of participant drinking 1ml water, the distance between hyoid and chin at rest minus distance during hyoid and chin are nerest. Repeated three times, and the mean value is further into analysis.

SECONDARY OUTCOMES:
SSA | Befor and after the three-week treatment, and 3 weeks after the treatment.
  Standardized swallowing assessment (SSA) include clinical examination, drinking 5mL water test and drinking 60mL water test.lowest score is 18, and the highest score is 46, high score indicationg poor condition.
FOIS | Befor and after the three-week treatment, and 3 weeks after the treatment.
  Functional oral intake scale. From one to seven, high score indicate better oral intake function.
DSRS | Befor and after the three-week treatment, and 3 weeks after the treatment.
  The Dysphagia Severity Rating Scale (DSRS) assigns a score to the feeding status achieved by the dysphagic patient depending on the categories of feeding stage for fluid and dietary consumption in addition to the level of dependency required for feeding. The score for each category can vary between 0 and 4 points, and is added to give a composite score. These scores were calculated by a speech and language therapist with special interest in neurogenic dysphagia. SALT：speech and language therapist.

OTHER OUTCOMES:
fNIRS | Befor and after the three-week treatment, and 3 weeks after the treatment.
  Functional near-infrared spectroscopy (fNIRS) is a tool for measuring the HbO2 concentration to reflect the excitation of cortex. Further analysis can help to explain the network of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Wang, professor, Principal Investigator — Qilu Hospital of Shandong University
Locations (2):
- China (2):
  - Qilu hospital of Shandong University, Jinan, Shandong
  - Yonghui Wang, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nowrin I, Bhattacharyya DS, Saif-Ur-Rahman KM. Community-based interventions to prevent stroke in low-income and middle-income countries: a protocol for a systematic review and meta-analysis. BMJ Open. 2022 Aug 8;12(8):e063181. doi: 10.1136/bmjopen-2022-063181. PMID 35940843
- [Background] Chiang CF, Lin MT, Hsiao MY, Yeh YC, Liang YC, Wang TG. Comparative Efficacy of Noninvasive Neurostimulation Therapies for Acute and Subacute Poststroke Dysphagia: A Systematic Review and Network Meta-analysis. Arch Phys Med Rehabil. 2019 Apr;100(4):739-750.e4. doi: 10.1016/j.apmr.2018.09.117. Epub 2018 Oct 21. PMID 30352222
- [Background] Palmer PM, McCulloch TM, Jaffe D, Neel AT. Effects of a sour bolus on the intramuscular electromyographic (EMG) activity of muscles in the submental region. Dysphagia. 2005 Summer;20(3):210-7. doi: 10.1007/s00455-005-0017-x. PMID 16362509